CLINICAL TRIAL: NCT01416376
Title: A Double Blind, Placebo Controlled, Phase I Dose-ranging Study to Evaluate the Activity of SRT2379 on Endotoxin Induced Inflammatory Response in Healthy Male Subjects
Brief Title: Effect of Multiple Dose Levels of SRT2379 on Endotoxin-Induced Inflammation
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Sirtris, a GSK Company (Industry)
Collaborators: GlaxoSmithKline (Industry)
Responsible Party: Sponsor
Organization: GlaxoSmithKline (Industry)
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Basic Science
Other Study IDs: 115830
Record Dates: First submitted 2011-07-28; First posted 2011-08-15 (Estimated); Last update posted 2017-06-15 (Actual); Status verified 2017-06

CONDITIONS: Sepsis
MeSH Terms: conditions — Sepsis

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (4):
- 50mg SRT2379 (Active Comparator): Single oral administration of 50mg SRT2379
  Interventions: Drug: Placebo
- 250mg SRT2379 (Active Comparator): Single oral administration of 250mg SRT2379
  Interventions: Drug: Placebo
- 1000mg SRT2379 (Active Comparator): Single oral administration of 1000mg SRT2379
  Interventions: Drug: SRT2379
- Placebo (Placebo Comparator): Single oral administration of placebo
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: SRT2379 — SRT2379 is supplied as hard gelatin capsules containing either 25mg or 250mg free-base equivalent of SRT23790 drug substance as its succinate salt.
  Arms: 1000mg SRT2379
Drug: Placebo — For the placebo capsules, the SRT2379 drug substance will be replaced by microcrystalline cellulose (Avicel PH200) to visually match the SRT2379 investigational product.
  Arms: 250mg SRT2379; 50mg SRT2379; Placebo

SUMMARY:
SRT2379 is a potent small molecule activator of SIRT1 that has been found to inhibit systemic inflammation induced by intravenous injection of lipopolysaccharide (LPS) in mice. The objective of this study is to determine the effect of a single administration of SRT2379, at multiple-dose levels, on the inflammatory response to low dose endotoxin.

ELIGIBILITY:
Inclusion Criteria:

* Healthy, as determined by a responsible and experienced physician, based on a medical evaluation including medical history, physical examination (PE) and laboratory tests carried out within 21 days prior to Day 1. A subject with a clinical abnormality or laboratory parameters outside the reference range for the population being studied may be included only if the Investigator and the Medical Monitor agree that the finding is unlikely to introduce additional risk factors and will not interfere with the study procedures
* Male between 18 and 35 years of age, inclusive, at the time of signing the informed consent
* Capable of giving written informed consent and able to comply with the requirements and restrictions listed in the informed consent form

  - Chemistry panel, including renal and liver function tests, without any clinically relevant abnormality as judged by the Investigator
* Subjects must agree to use double-barrier birth control or abstinence while participating in the study and for 7 days following the last dose of study drug

Exclusion Criteria:

* Subject has had a major illness in the past 3 months or any significant chronic medical illness that the Investigator would deem unfavourable for enrolment, including inflammatory diseases
* Subjects with a history of any type of malignancy with the exception of successfully treated basal cell cancer of the skin
* Subject has a past or current gastrointestinal disease which may influence drug absorption
* The subject has a known positive test for hepatitis C antibody, hepatitis B surface antigen or human immunodeficiency virus (HIV) antibody 1 or 2

  * Current or chronic history of liver disease, or known hepatic or biliary abnormalities (with the exception of Gilbert's syndrome or asymptomatic gallstones)
  * Subject has a history, within 3 years, of drug abuse (including benzodiazepines, opioids, amphetamine, cocaine, THC, methamphetamine) or a positive drug result at the Screening visit
  * History of alcoholism and/or is drinking more than 3 units of alcohol per day. Alcoholism is defined as an average weekly intake of >21 units for males. One unit is equivalent to 8 g of alcohol: a half-pint (~240 mL) of beer, 1 glass (125 mL) of wine or 1 (25 mL) measure of spirits
  * The subject has received an investigational product within three months of the first dosing day in the current study; Note: any subject who has participated in a prior human endotoxemia study with SRT2379 or SRT2104 would be excluded from participation in this trial.
  * Use of prescription or non-prescription drugs and herbal and dietary supplements within 7 days unless in the opinion of the Investigator the medication will not interfere with the study procedures or compromise subject safety
  * Subject has difficulty donating blood or limited accessibility of a vein in left and right arm
* Subject has donated more than 350 mL of blood in last 3 months
* Subject uses tobacco products

  * Any clinically relevant abnormality noted on the 12-lead ECG as judged by the Investigator or an average QTcB or QTcF > 450 msec
  * Any other issue that, in the opinion of the Investigator , could be harmful to the subject or compromise interpretation of the data
* Prior participation in a trial where the subject received intravenous endotoxin (LPS) infusion

Ages: 18 Years to 35 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 39 (Actual)
Dates: Start 2011-08-30 (Actual); Primary Completion 2011-12-12 (Actual); Study Completion 2011-12-12 (Actual)

PRIMARY OUTCOMES:
Clinical signs and symptoms of inflammation will be used as a measure of the effect of multiple-dose levels of SRT2379 on the inflammatory response in normal healthy male subjects exposed to low-dose endotoxin (LPS). | 12 days
Laboratory parameters of inflammation will be used as a measure of the effect of multiple-dose levels of SRT2379 on the inflammatory response in normal healthy male subjects exposed to low-dose endotoxin (LPS). | 12 days

SECONDARY OUTCOMES:
Plasma levels of SRT2379 will be measured to assess the pharmacokinetics of SRT2379 in healthy male subjects exposed to low-dose endotoxin (LPS). | 2 days
Number of participants with adverse events and incidence of adverse events will be used as a measure of safety and tolerability of multiple-dose levels of SRT2379 in healthy male subjects exposed to low-dose endotoxin (LPS). | 34 days

CONTACTS AND LOCATIONS:
Overall Officials: GSK Clinical Trials, Study Director — GlaxoSmithKline
Locations (1):
- GSK Investigational Site, Amsterdam, Netherlands

IPD SHARING:
Plan to Share IPD: Yes
Patient-level data for this study will be made available through www.clinicalstudydatarequest.com following the timelines and process described on this site.

REFERENCES:
- See also: Results for study 115830 can be found on the GSK Clinical Study Register. — https://www.gsk-clinicalstudyregister.com/study/115830?search=study&search_terms=115830#rs
- See also: Researchers can use this site to request access to anonymised patient level data and/or supporting documents from clinical studies to conduct further research. — https://www.clinicalstudydatarequest.com
- Available data/document: Clinical Study Report: 115830 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Dataset Specification: 115830 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Individual Participant Data Set: 115830 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Statistical Analysis Plan: 115830 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Study Protocol: 115830 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Informed Consent Form: 115830 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register